CLINICAL TRIAL: NCT00116298
Title: A Study to Compare Long-Term Safety and Tolerability of Stavudine (d4T) Extended Release (ER) Versus Conventional (Immediate Release, IR) Formulations, Each In Combination With Lamivudine (3TC) and Efavirenz (EFV) in Subjects Who Have Completed BMS Studies AI455-096 and AI455-099
Brief Title: Rollover Study for Zerit (Stavudine) ER Studies (-096, -099)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI455-110
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections; AIDS
Keywords: Antivirals; HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Stavudine; efavirenz; Lamivudine

INTERVENTIONS:
Drug: stavudine, efavirenz, lamivudine

SUMMARY:
The purpose of this study is to compare long-term safety and tolerability of stavudine (d4T) extended release (ER) versus conventional (immediate release [IR]) formulations, each in combination with lamivudine (3TC) and efavirenz (EFV) in subjects who have completed Bristol-Myers Squibb (BMS) studies AI455-096 and AI455-099.

ELIGIBILITY:
Inclusion Criteria:

* Completed d4T studies AI455-096 or AI455-099
* Have demonstrated compliance with the study medication and treatment visits
* Provide written informed consent
* Agree to use a barrier method of birth control (such as condoms) during the study
* Have a negative pregnancy test within 72 hours prior to start of study medication

Exclusion Criteria:

* Are pregnant or breast-feeding
* Need to take certain medications that have systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic or cytotoxic potential
* Have active alcohol or substance abuse which may prevent compliance or increase risk of developing pancreatitis
* Have certain other conditions or prior treatments that might interfere with study continuation
* Need to take certain medications that should not be taken with EFV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 2001-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Safety: Frequency and severity of AEs, and treatment discontinuations for AEs; population trends for triglycerides and cholesterol. Primary efficacy outcome: proportion of subjects with HIVRNA <400, <50, and change in viral load over the study period

SECONDARY OUTCOMES:
Efficacy: Changes in CD4 cell counts

CONTACTS AND LOCATIONS:
Locations (63):
- United States (19):
  - Local Institution, Berkeley, California
  - Local Institution, Los Angeles, California
  - Local Institution, West Hollywood, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Brookline, Massachusetts
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Reno, Nevada
  - Local Institution, New York, New York
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Hampton, Virginia
- Argentina (4):
  - Local Institution, San Isidro, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
  - Local Institution, Córdoba
- Belgium (2):
  - Local Institution, Ghent
  - Local Institution, Liège
- Brazil (4):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Belo Horizonte - MG, Minas Gerais
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Santos, São Paulo
- Canada (3):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- France (5):
  - Local Institution, Bordeaux
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Rennes
- Israel (2):
  - Local Institution, Rehovot
  - Local Institution, Tel Hashorner
- Italy (7):
  - Local Institution, Bari
  - Local Institution, Bergamo
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Pisa
  - Local Institution, Torino
- Local Institution, Mexico City, Mexico City, Mexico
- Portugal (2):
  - Local Institution, Coimbra
  - Local Institution, Lisbon
- Puerto Rico (2):
  - Local Institution, Cotto Laurel
  - Local Institution, San Juan
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (5):
  - Local Institution, Bedford Gardens, Gauteng
  - Local Institution, Hatfield, Gauteng
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Westdene, Gauteng
  - Local Institution, Tygerberg, Western Cape
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Nontaburi